CLINICAL TRIAL: NCT00036309
Title: Duloxetine Versus Placebo in the Prevention of Relapse of Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Purpose: Treatment
Other Study IDs: 4445; F1J-MC-HMBC
Record Dates: First submitted 2002-05-08; First posted 2002-05-09 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Depressive Disorder
Keywords: Major Depressive Disorder; Diagnostic and Statistical Manual of Mental Disorders Fourth Edition-defined major depressive disorder without psychotic features
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Disease | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine Hydrochloride

SUMMARY:
The purpose of this study is to determine if duloxetine is effective when compared to placebo in preventing recurrence of major depressive disorder in patients who have responded to open-label duloxetine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent
* Meet criteria for major depressive disorder without psychotic features.
* Have a level of understanding sufficient to provide informed consent and to communicate with the investigator and site personnel.
* Have had at least one other major depressive episode prior to the one being experienced at study entry.
* You are reliable and agree to keep all appointments for clinic visits, tests and procedures required by the protocol.

Exclusion Criteria:

* You have had treatment with a drug within the last 30 days that has not received regulatory approval at the time of study entry.
* Any women who are pregnant or breast feeding.
* If you have any serious medical illnesses other than major depressive disorder.
* If you have previously participated in a clinical trial for duloxetine.
* Any previous or current diagnosis of bipolar, schizophrenia, or other psychotic disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-05; Study Completion 2003-07

CONTACTS AND LOCATIONS:
Locations (1):
- For information on a site near you, call our call center at 1-877-CTLILLY (1-877-285-4559), Durham, North Carolina, United States

REFERENCES:
- [Derived] Hudson JI, Perahia DG, Gilaberte I, Wang F, Watkin JG, Detke MJ. Duloxetine in the treatment of major depressive disorder: an open-label study. BMC Psychiatry. 2007 Aug 28;7:43. doi: 10.1186/1471-244X-7-43. PMID 17725843